CLINICAL TRIAL: NCT04140539
Title: A Single Arm, Open Label Clinical Study to Enable Process Validation of Commercial Grade Ex Vivo Hematopoietic Stem Cell Gene Therapy (OTL-101) in Subjects With Severe Combined Immunodeficiency Due to Adenosine Deaminase Deficiency (ADA-SCID)
Brief Title: A Clinical Study to Enable Process Validation of Commercial Grade OTL-101
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment on hold for business reasons. Study will not be performed.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Donald B. Kohn, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTL-101-7
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Severe Combined Immunodeficiency Due to ADA Deficiency
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gene Therapy (Experimental): Infusion OTL-101
  Interventions: Biological: OTL-101

INTERVENTIONS:
Biological: OTL-101 — Autologous CD34+ cell enriched population that contains hematopoietic stem and progenitor cells (HSPCs) transduced ex vivo using a lentiviral vector (LV) encoding the human adenosine deaminase (ADA) gene.

SUMMARY:
The purpose of the current study is to treat at least 3 ADA-SCID patients with OTL-101 prepared by the commercial manufacturing process.

DETAILED DESCRIPTION:
The safety and efficacy of OTL-101 for the treatment of patients with ADA- SCID have been established in previous clinical trials. The purpose of the current study is to treat at least 3 ADA-SCID patients with OTL-101 prepared by the commercial manufacturing process in order to facilitate collection of data necessary for final manufacturing.

Assessments will focus on monitoring safety and engraftment, through the evaluation of parameters describing immunological recovery, ADA enzyme activity and persistence of gene marking (VCN) at 6 months and 12 months. After completion of 12 months of follow-up on the current study protocol, subjects will be enrolled in an observational long-term follow-up study, in order to monitor the long-term safety of treatment with OTL-101.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent by the subject or parent(s)/legal guardian(s), prior to any study related procedures taking place. Where consent is provided by the parent(s)/legal guardian(s), assent by the subject should also be sought, if appropriate
* Age ≥30 days and <18 years
* Diagnosis of ADA-SCID based on either:

  * 1) Evidence of ADA deficiency, defined as Decreased ADA enzymatic activity in erythrocytes, leukocytes, skin fibroblasts, or in cultured fetal cells to levels consistent with ADA-SCID as determined by the reference laboratory OR Identified mutations in ADA alleles consistent with a severe reduction in ADA activity
  * 2) Evidence of ADA-SCID, defined as Family history of a first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency OR Evidence of severe immunologic deficiency in subjects prior to the institution of immune restorative therapy, based on at least one of the following:

    * Lymphopenia (absolute lymphocyte count <400 cells/μL) OR absence or low number of T cells (absolute CD3+ count < 300 cells/μL)
    * Severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (either <10% of lower limit of normal controls for the diagnostic laboratory, or <10% of the response of the normal control of the day, or stimulation index <10)
    * Identification of SCID by neonatal screening revealing low T cell receptor excision circles (TREC) levels
* Ineligible for allogeneic bone marrow transplantation from an Human leukocyte antigen (HLA)-identical sibling donor, with normal immune function
* For females of child-bearing potential, negative pregnancy test up to 30 days prior to the Screening visit. For all subjects in the reproductive age range, agreement to use highly effective and adequate method of contraception while receiving treatment and for at least 12 months following drug administration
* Willingness and ability of the subjects and parent(s)/legal guardian(s) to comply with study procedures and requirements, including remaining at the clinic for the required duration of conditioning and treatment and compliance with follow-up evaluations

Exclusion Criteria:

* Ineligible for autologous HSCT as per clinical site criteria.
* Hematologic abnormality, defined as:

  * Anemia (Hb <8.0 g/dL)
  * Neutropenia (absolute neutrophil count (ANC) <500 cells/mm3). Note: ANC <500 cells/mm3 with absence of myelodysplastic syndrome on bone marrow aspirate and biopsy and normal marrow cytogenetics are acceptable for eligibility
  * Thrombocytopenia (platelet count <50,000 platelets/mm3)
  * Prothrombin Time (PT) or International Normalized Ratio (INR) and Partial thromboplastin time (PTT) >2 times the upper limit of normal (ULN) (subjects with a correctable deficiency controlled on medication will not be excluded)
  * Cytogenetic abnormalities on peripheral blood or bone marrow or amniotic fluid (if available)
  * Prior allogeneic HSCT with cytoreductive conditioning
* Pulmonary abnormality, defined as:

  * Resting oxygen (O2) saturation by pulse oximetry <90% on room air
  * Chest X-ray indicating active or progressive pulmonary disease. Note: Chest X- ray indicating residual signs of treated pneumonitis is acceptable for eligibility
* Cardiac abnormality, defined as:

  * Abnormal electrocardiogram indicating cardiac pathology
  * Uncorrected congenital cardiac malformation with clinical symptoms
  * Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension
  * Poor cardiac function as evidenced by left ventricular ejection fraction <40% on echocardiogram
* Neurologic abnormality, defined as:

  * Significant neurologic abnormality revealed by examination
  * Uncontrolled seizure disorder
* Renal abnormality, defined as:

  * Renal insufficiency: serum creatinine ≥1.2 mg/dL (106 μmol/L), or ≥3+ proteinuria
  * Abnormal serum sodium, potassium, calcium, magnesium or phosphate levels at >2 times the ULN
* Hepatic/gastrointestinal abnormality, defined as:

  * Serum transaminases >5 times the ULN
  * Serum bilirubin >2 times the ULN
  * Serum glucose >1.5 times the ULN
* Oncologic disease, defined as:

  * Evidence of active malignant disease other than Dermatofibrosarcoma protuberans (DFSP)
  * Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells (if anti-neoplastic therapy has been completed, a subject with a history of DFSP can be included)
  * Evidence of DFSP expected to be life limiting within the 5 years following the infusion of genetically corrected cells
* Known sensitivity to busulfan
* Confirmation of infectious disease at time of Screening assessment for:

  * Human Immunodeficiency Virus (HIV)-1 and HIV-2
  * Hepatitis B and Hepatitis C
  * Parvovirus B19
  * Human T-cell lymphotropic virus (HTLV)-1 and HTLV-2
* Pregnant at the time of Screening
* Affected by a major congenital anomaly
* Likely to require treatment during the study with drugs that are not permitted by the study protocol
* Previously treated with another form of gene therapy
* Affected by any other condition(s) which, in the opinion of the Principal Investigator, contraindicate bone marrow harvest, the administration of busulfan and the infusion of OTL-101, or which indicate an inability of the subject or subject's parent(s)/legal guardian(s) to comply with the protocol

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Adenosine Deaminase (ADA) enzyme activity | 6 months post treatment
  ADA enzyme activity in red blood cells
T cell (CD3+) count | 6 months post treatment
  Absolute count of CD3+ cells
Vector Copy Number (VCN) | 6 months post treatment
  VCN in granulocytes

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months post treatment
  OS will be defined as the proportion of subjects alive at 12 months post-treatment with OTL-101
Event-free Survival (EvFS) | 12 months post treatment
  EvFS will be defined as the proportion of subjects alive with no "event", an event being the resumption of Pegylated adenosine deaminase (PEG-ADA) Enzyme Replacement Therapy (ERT) or the need for a rescue allogeneic hematopoietic stem cell transplant (HSCT) at 12 months post-treatment with OTL-101

CONTACTS AND LOCATIONS:
Overall Officials: Orchard Therapeutics Clinical Trials, Study Director — Orchard Therapeutics (Europe) Limited
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No